CLINICAL TRIAL: NCT02062879
Title: Ketamine Patient-Controlled Analgesia for Acute Pain in Native Airway Multiple and Orthopedic Trauma Patients: A Randomized, Active Comparator, Blinded Trial
Brief Title: Ketamine Patient-Controlled Analgesia for Acute Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawals from study due to anticipated effects from study drugs
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Sheila Takieddine, Policy Development Specialist, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mueller2014
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Acute Pain; Multiple Trauma; Fractures
Keywords: pain; trauma
MeSH Terms: conditions — Acute Pain; Multiple Trauma; Fractures, Bone; Pain; Wounds and Injuries | interventions — Ketamine; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Ketamine 90mg/30 mL PCA (3 mg/mL)
  Interventions: Drug: Ketamine
- Hydromorphone (Active Comparator): Hydromorphone 6mg/30 mL PCA (0.2 mg/mL)
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Ketamine — Ketamine administered as patient-controlled analgesia.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Hydromorphone — Hydromorphone administered as patient-controlled analgesia.
  Other Names: Dilaudid
  Arms: Hydromorphone

SUMMARY:
This study will compare ketamine and hydromorphone as alternative patient-controlled interventions for trauma-related pain. Patients receiving ketamine PCA are expected to require less total and breakthrough opioid and to have similar or improved objective pain scores. Patients receiving ketamine are also expected to have shorter duration of supplemental oxygen requirement, fewer episodes of oxygen desaturation, improved pulmonary toilet, lower use of antiemetics, and shorter times to first bowel movement. Ketamine is further expected to be associated with decreased intensive care unit and hospital lengths of stay, faster time to maximum allowable ambulation, decreased opioid dosage at discharge, and lower report of chronic pain syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Total Injury Severity Score greater than 9
* Functioning intravenous catheter present per standard of care
* Patient planned to receive PCA for acute pain per standard of care
* Patient ability to effectively use a PCA device as assessed by the primary attending trauma service
* Negative pregnancy test for women of childbearing age

Exclusion Criteria:

* Body mass index greater than 35
* History of active psychiatric disease
* Acute or chronic liver or renal failure
* History of heart failure or coronary artery disease
* Patients with documented chronic pain syndrome who use opioids as maintenance medication in outpatient therapy
* Patients who abuse alcohol and are at high risk for alcohol withdrawal
* Intubated patients
* Glasgow Coma Scale score less than 13, or motor subscore less than 6
* Documented allergy to ketamine, hydromorphone, or lorazepam
* Pregnancy
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila C Takieddine, Pharm.D., Principal Investigator — UC Health; Eric W Mueller, Pharm.D., Principal Investigator — UC Health
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Takieddine SC, Droege CA, Ernst N, Droege ME, Webb M, Branson RD, Gerlach TW, Robinson BRH, Johannigman JA, Mueller EW. Ketamine versus hydromorphone patient-controlled analgesia for acute pain in trauma patients. J Surg Res. 2018 May;225:6-14. doi: 10.1016/j.jss.2017.12.019. Epub 2018 Jan 8. PMID 29605036

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Hydromorphone
Started | 10 | 10
Completed | 6 | 9
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Hydromorphone | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [28 to 47] | 26 [22 to 30] | 30 [25 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 27 [23.8 to 29] | 26.5 [21.7 to 29] | 27 [23 to 29]
Injury Severity Score [Median (Inter-Quartile Range); unit: scores on a scale] — The Injury Severity Score is an anatomical scoring system that correlates with morbidity and mortality. The value can range from 0 to 75. Higher values represent a worse outcome. Reference: Baker SP et al, "The Injury Severity Score: a method for describing patients with multiple injuries and evaluating emergency care", J Trauma 14:187-196;1974.
  scores on a scale | 29 [22 to 33] | 28 [26 to 29] | 29 [26 to 29]
Blunt Trauma [Count of Participants; unit: Participants] | 10 | 9 | 19
Penetrating Trauma [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Daily Opioid Requirement
Description: Daily breakthrough opioid requirement plus non-breakthrough opioid use in milligrams of morphine equivalents
Time Frame: Participants will be followed for their entire hospital stay, an expected average of 1 week.
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalents/day
Arm/Group | Ketamine | Hydromorphone
Number analyzed (Participants) | 10 | 10
mg morphine equivalents/day | 10 [4.2 to 15] | 42.5 [31.7 to 62]

2. Secondary Outcome: Breakthrough Daily Opioid Requirement
Description: Breakthrough daily opioid requirement in milligrams of morphine equivalents/day
Time Frame: Participants will be followed for their entire hospital stay, an expected average of 1 week
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalents/day
Arm/Group | Ketamine | Hydromorphone
Number analyzed (Participants) | 10 | 10
mg morphine equivalents/day | 10 [0.63 to 19.38] | 10 [4.38 to 22.5]

3. Secondary Outcome: Median Pain Score
Description: Median daily pain score measures on a visual analogue scale for pain, with a range of 0 to 10. Higher scored indicate worse pain.
Time Frame: Participants will be followed for their entire hospital stay, an expected average of 1 week
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Ketamine | Hydromorphone
Number analyzed (Participants) | 10 | 10
scores on a scale | 6.3 [4 to 7.5] | 5.3 [3 to 6.8]

ADVERSE EVENTS:
Arm/Group | Ketamine | Hydromorphone
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 7/10 | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=10) | Hydromorphone (N=10)
Hallucinations (Psychiatric disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 5 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No